CLINICAL TRIAL: NCT01729299
Title: Ghrelin Effect on Beta Cell Function in Health and Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: David Dalessio (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, David Dalessio, Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 12070904
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes
Keywords: ghrelin; glucose control; GLP-1; Exendin (9-39); insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — exendin (9-39); acyl-ghrelin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- saline (Placebo Comparator): Saline: 0.9% saline solution
  Interventions: Drug: saline
- ghrelin and exendin (9-39) (Experimental): Ghrelin+Ex-9: Combination of ghrelin and Ex-9,
  Interventions: Drug: Exendin (9-39); Drug: acyl ghrelin
- Exendin (9-39) (Experimental): Exendin (9-39) (25 µg/kg) bolus over 1 min followed by a continuous infusion of 2.5 µg/kg/min
  Interventions: Drug: Exendin (9-39)
- ghrelin (Experimental): synthetic human Acyl Ghrelin (0.28 μg/kg) bolus over 1 min followed by 2 μg/kg/h continuous infusion,
  Interventions: Drug: acyl ghrelin

INTERVENTIONS:
Drug: Exendin (9-39)
  Arms: Exendin (9-39); ghrelin and exendin (9-39)
Drug: acyl ghrelin
  Arms: ghrelin; ghrelin and exendin (9-39)
Drug: saline
  Arms: saline

SUMMARY:
To determine the role of nutrient status on ghrelin regulation of insulin secretion. We hypothesize that ghrelin and glucagon-like peptide-1 (GLP-1)(both are hormones made in the gut,) have differential effects on β-cell function in the fed state. We will compare insulin secretion and glucose turnover during meal ingestion using a dual glucose tracer and mixed meal protocol in subjects receiving ghrelin or saline. We will also determine the role of ghrelin-stimulated GLP-1 levels in this process using the GLP-1 receptor (GLP-1R) antagonist Exendin(9-39) (Ex-9).

DETAILED DESCRIPTION:
We plan to study 20 healthy subjects on 4 occasions where they will receive ghrelin, ghrelin+Ex-9, Ex-9 or saline infusion after an overnight fast in a randomized order; Ex-9 will be used to block GLP-1 action. A 240-minute meal tolerance test (MTT) using a dual glucose tracer method will serve as the foundation of each study visit. One tracer, [6,6-2H2]glucose will be infused intravenously before and during the test meal to quantify fasting endogenous glucose production (EGP), and glucose disappearance during the meal. A second tracer, [U-13C]glucose, will be included in the meal to trace the appearance of oral glucose. The systemic appearance rates of both ingested tracer and total (i.e., ingested and endogenously produced) glucose will be calculated. Using this protocol, we will be able to evaluate a) insulin secretion in response to mixed-meal ingestion, b) glucose appearance and glucose disappearance during meal ingestion, c) the ghrelin effect on these parameters without GLP-1, and d) the effect of GLP-1 in the response based on the effects with and without Ex-9.

This dual-tracer method has been used to assess the ability of an individual to dispose of an oral glucose load, and accurately fractionates the appearance of ingested glucose in plasma (Ra meal), EGP, and peripheral glucose disposal (Rd) in this setting 41-42. The [6,6-2H2]glucose and [U-13C]glucose are stable-isotope tracers and are different from radioactive-isotope tracers in that they do not emit radiation.

All procedures will be performed at the CTRC at the Cincinnati Children's Hospital Medical Center (CCHMC).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women
2. Ages between 18 and 45 years
3. BMI between 18 and 29 kg/m2

Exclusion Criteria:

1. History or clinical evidence of impaired fasting glucose or diabetes mellitus, myocardial infarction within the past year, history or symptoms of congestive heart failure, uncontrolled hypertension, history or active liver or renal disease (AST or ALT >2x upper limits of normal, calculated glomerular filtration rate [GFR] <60).
2. History of pituitary or adrenal disorders or neuroendocrine tumor.
3. Anemia defined as hematocrit <33%.
4. Use of medications that alter glucose metabolism
5. Pregnancy or lactation.
6. Abnormal Electrocardiogram (ECG): evidence of ischemia or arrhythmia.
7. Women who have a positive pregnancy test at any time during the study period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
post-prandial insulin secretion | 1 year
  Postprandial insulin secretion (ISR-meal) will be derived from plasma C-peptide concentrations during MTT using deconvolution with population estimates of C-peptide clearance.

SECONDARY OUTCOMES:
endogenous GLP-1 contribution to postprandial insulin secretion | 1 year
  The endogenous GLP-1 contribution to postprandial insulin secretion (GLP-1 effect) will be calculated as the difference in ISR-meal with and without Ex-9.
β-cell response to glucose | 1 year
  An index of β-cell response to glucose will be calculated as the incremental insulin/glucose (I/G) AUC (ΔAUCI/G).
insulin sensitivity | 1 year
  Whole body insulin sensitivity will be estimated using the Matsuda Index that has been well validated in large cohort studies and has demonstrated a good correlation with IVGTT or hyperinsulinemic-euglycemic clamp derived measures of insulin sensitivity. β-cell function (DI-meal) will be calculated as ΔAUCI/G x Matsuda Index
fasting EGP | 1 year
  Fasting EGP will be calculated as the ratio of 6,6-[2H2]glucose infusion rate to plasma tracer enrichment (tracer-to-tracee ratio [TTR]6,6 from measurements obtained in the last 20 min of the basal tracer equilibration period, when plasma glucose concentration and 6,6-[2H2]glucose enrichment are stable).
glucose appearance | 1 year
  Total rates of glucose appearance after meal ingestion (total Ra) will be calculated by modeling 6,6-[2H2] enrichment ([TTR]6,6) using both a two-compartment model and Steele's equation42. Meal glucose appearance will be determined from the analysis of [U-13C]-glucose fluxes. The meal will be labeled to 2.66% with U-13C]-glucose (TTRmeal). From the measurement of plasma [TTR]13C, we will calculate the exogenous (meal) glucose concentrations, [Gmeal] , from total glucose concentrations, [Gtot] , using the formula [Gmeal] = [Gtot] x [TTR]13C / TTRmeal as previously described 42,45. Endogenous glucose concentration [Gend] will be calculated as [Gend] = [Gtot] - [Gmeal].
EGP during MTT | 1 year
  EGP during MTT will be calculated using model analysis of TTR of endogenous glucose ([TTR]end) and calculated as [TTR]end = [TTR]6,6 x [Gtot] / [Gend]
exogenous glucose rate of appearance | 1 year
  Exogenous glucose rate of appearance, Ra meal, will be calculated by subtracting EGP during meal from total Ra (Ra meal = total Ra - EGP).
metabolic glucose clearance | 1 year
  As for indexes of peripheral insulin sensitivity, we will calculate metabolic glucose clearance during MTT using peripheral glucose disposal (Rd) divided by glucose concentration (expressed as ml/min/kg) where Rd is calculated by subtracting the rate of change of plasma glucose mass from total Ra.
area under the curve | 1 year
  AUC for glucagon, GLP-1, GIP, and free fatty acids (FFA), a measure of lipolysis.
ghrelin measures | 1 year
  AG and total ghrelin levels will be measured during clamp-MTT.
gastric emptying | 1 year
  Gastric emptying estimated by the gastric half-emptying time calculated from the emptying curve as the time when 50% of the total cumulated dose of acetaminophen has been eliminated46.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Tong, MD, MPH, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Page LC, Gastaldelli A, Gray SM, D'Alessio DA, Tong J. Interaction of GLP-1 and Ghrelin on Glucose Tolerance in Healthy Humans. Diabetes. 2018 Oct;67(10):1976-1985. doi: 10.2337/db18-0451. Epub 2018 Jul 31. PMID 30065032